CLINICAL TRIAL: NCT05348109
Title: Assessment of Decision Support System Software in Extraction and Anchorage Planning Among Adult Patients Using Computer Algorithm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Walaa Mohamed Hassan Gadallah, Orthodontics Master candidate, Cairo University
Other Study IDs: 94030405
Record Dates: First submitted 2021-12-21; First posted 2022-04-27 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Cases That Need Extraction of Teeth in Orthodontics; Anchorage Planning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- well fininshed cases
  Interventions: Other: Well finished cases

INTERVENTIONS:
Other: Well finished cases — To decide whether extraction or non-extraction decision will be made for each case
  Other Names: extraction and non-extraction in well finished cases

SUMMARY:
It was introduced in dentistry to be used in innovative research and development in addition to facilitating the decision in complicated cases and ensure high patient care quality. In the field of Orthodontics in specific, many studies previously mentioned the idea of artificial intelligence showing very promising results and high degree of reliability. It was used in different domains in orthodontics like diagnosis, treatment planning, evaluation of treatment outcome

DETAILED DESCRIPTION:
In this study, the aim is to access the efficiency of the new decision support system in determining whether the decision is extraction or non-extraction and the anchorage plan required for each case. This was performed in the past in many countries and those studies are published

ELIGIBILITY:
Inclusion Criteria:

1. Cases with well finished orthodontic treatment.
2. Cases with history of crowding more than 10 mm and requiring extraction.
3. Cases with no severe skeletal discrepancy.
4. Well documented cases with both pre-operative and post-operative records.
5. Patients with a full set of permanent teeth erupted

Exclusion Criteria:

1. Improperly finished orthodontic cases.
2. Cases with mild crowding managed by treatment options other than extraction.
3. Growing patients or showing any residual growth remaining in cephalometric analysis
4. Cases with severe skeletal discrepancy.
5. Poorly documented cases.
6. Patients not sticking to anchorage plan

Ages: 15 Years to 35 Years | Sex: All
Age Groups: Child, Adult
Study Population: Recruiting well finished cases having history of crowding from Kasr el Ainy with no severe skeletal discrepancy, cases should be well documented. The precise and complete documentation of the patients in terms of the presence of:
  1. Preoperative and postoperative x-rays.
  2. Good quality preoperative and postoperative photographs.
  3. Preoperative and postoperative study models.
  4. Detailed documentation of the treatment sequence and mechanics. If there were incomplete data provided in the patient's file; the patient will then be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-08-22 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
To study the efficiency of the program decisions in terms of extraction/non-extraction and Anchorage planning decisions | 1 year
  The concordance correlation coefficient would be used to measure the agreement between the 2 methods on the basis of the values (%) assigned for each treatment option by the 2 methods (quantitative data).

CONTACTS AND LOCATIONS:
Locations (1):
- Walaa Mohamed Hassan Gadallah, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mandava, P., Ganugapanta, V. R. and Pradesh, A. (2016) 'Review article Annals and Essences of Dentistry ANCHORAGE IN ORTHODONTICS : A LITERATURE REVIEW Review article', Annals and Essences of Dentistry, VIII(2).
- [Background] Muraev AA, Tsai P, Kibardin I, Oborotistov N, Shirayeva T, Ivanov S, Ivanov S, Guseynov N, Aleshina O, Bosykh Y, Safyanova E, Andreischev A, Rudoman S, Dolgalev A, Matyuta M, Karagodsky V, Tuturov N. Frontal cephalometric landmarking: humans vs artificial neural networks. Int J Comput Dent. 2020;23(2):139-148. PMID 32555767
- [Result] Aksakalli S, Demir A, Selek M, Tasdemir S. Temperature increase during orthodontic bonding with different curing units using an infrared camera. Acta Odontol Scand. 2014 Jan;72(1):36-41. doi: 10.3109/00016357.2013.794954. Epub 2013 May 3. PMID 23638766
- [Result] Auconi P, Scazzocchio M, Cozza P, McNamara JA Jr, Franchi L. Prediction of Class III treatment outcomes through orthodontic data mining. Eur J Orthod. 2015 Jun;37(3):257-67. doi: 10.1093/ejo/cju038. Epub 2014 Sep 4. PMID 25190642
- [Result] Bichu YM, Hansa I, Bichu AY, Premjani P, Flores-Mir C, Vaid NR. Applications of artificial intelligence and machine learning in orthodontics: a scoping review. Prog Orthod. 2021 Jul 5;22(1):18. doi: 10.1186/s40510-021-00361-9. PMID 34219198
- [Result] Briganti G, Le Moine O. Artificial Intelligence in Medicine: Today and Tomorrow. Front Med (Lausanne). 2020 Feb 5;7:27. doi: 10.3389/fmed.2020.00027. eCollection 2020. PMID 32118012
- [Result] Chen S, Wang L, Li G, Wu TH, Diachina S, Tejera B, Kwon JJ, Lin FC, Lee YT, Xu T, Shen D, Ko CC. Machine learning in orthodontics: Introducing a 3D auto-segmentation and auto-landmark finder of CBCT images to assess maxillary constriction in unilateral impacted canine patients. Angle Orthod. 2020 Jan;90(1):77-84. doi: 10.2319/012919-59.1. Epub 2019 Aug 12. PMID 31403836
- [Result] Chen YW, Stanley K, Att W. Artificial intelligence in dentistry: current applications and future perspectives. Quintessence Int. 2020;51(3):248-257. doi: 10.3290/j.qi.a43952. PMID 32020135
- [Result] Choi HI, Jung SK, Baek SH, Lim WH, Ahn SJ, Yang IH, Kim TW. Artificial Intelligent Model With Neural Network Machine Learning for the Diagnosis of Orthognathic Surgery. J Craniofac Surg. 2019 Oct;30(7):1986-1989. doi: 10.1097/SCS.0000000000005650. PMID 31205280
- [Result] Dorsey ER, Glidden AM, Holloway MR, Birbeck GL, Schwamm LH. Teleneurology and mobile technologies: the future of neurological care. Nat Rev Neurol. 2018 May;14(5):285-297. doi: 10.1038/nrneurol.2018.31. Epub 2018 Apr 6. PMID 29623949
- [Result] Felfoul O, Mohammadi M, Taherkhani S, de Lanauze D, Zhong Xu Y, Loghin D, Essa S, Jancik S, Houle D, Lafleur M, Gaboury L, Tabrizian M, Kaou N, Atkin M, Vuong T, Batist G, Beauchemin N, Radzioch D, Martel S. Magneto-aerotactic bacteria deliver drug-containing nanoliposomes to tumour hypoxic regions. Nat Nanotechnol. 2016 Nov;11(11):941-947. doi: 10.1038/nnano.2016.137. Epub 2016 Aug 15. PMID 27525475
- [Result] Feres M, Louzoun Y, Haber S, Faveri M, Figueiredo LC, Levin L. Support vector machine-based differentiation between aggressive and chronic periodontitis using microbial profiles. Int Dent J. 2018 Feb;68(1):39-46. doi: 10.1111/idj.12326. Epub 2017 Aug 2. PMID 28771699
- [Result] Goto S, Kimura M, Katsumata Y, Goto S, Kamatani T, Ichihara G, Ko S, Sasaki J, Fukuda K, Sano M. Artificial intelligence to predict needs for urgent revascularization from 12-leads electrocardiography in emergency patients. PLoS One. 2019 Jan 9;14(1):e0210103. doi: 10.1371/journal.pone.0210103. eCollection 2019. PMID 30625197
- [Result] Hamet P, Tremblay J. Artificial intelligence in medicine. Metabolism. 2017 Apr;69S:S36-S40. doi: 10.1016/j.metabol.2017.01.011. Epub 2017 Jan 11. PMID 28126242
- [Result] Hwang JJ, Lee JH, Han SS, Kim YH, Jeong HG, Choi YJ, Park W. Strut analysis for osteoporosis detection model using dental panoramic radiography. Dentomaxillofac Radiol. 2017 Oct;46(7):20170006. doi: 10.1259/dmfr.20170006. Epub 2017 Jul 14. PMID 28707523
- [Result] Khanagar SB, Al-Ehaideb A, Vishwanathaiah S, Maganur PC, Patil S, Naik S, Baeshen HA, Sarode SS. Scope and performance of artificial intelligence technology in orthodontic diagnosis, treatment planning, and clinical decision-making - A systematic review. J Dent Sci. 2021 Jan;16(1):482-492. doi: 10.1016/j.jds.2020.05.022. Epub 2020 Jun 5. PMID 33384838
- [Result] Kunz F, Stellzig-Eisenhauer A, Zeman F, Boldt J. Artificial intelligence in orthodontics : Evaluation of a fully automated cephalometric analysis using a customized convolutional neural network. J Orofac Orthop. 2020 Jan;81(1):52-68. doi: 10.1007/s00056-019-00203-8. Epub 2019 Dec 18. PMID 31853586
- [Result] Yeom SH, Na JS, Jung HD, Cho HJ, Choi YJ, Lee JS. Computational analysis of airflow dynamics for predicting collapsible sites in the upper airways: machine learning approach. J Appl Physiol (1985). 2019 Oct 1;127(4):959-973. doi: 10.1152/japplphysiol.01033.2018. Epub 2019 Jul 18. PMID 31318618
- [Result] Xie X, Wang L, Wang A. Artificial neural network modeling for deciding if extractions are necessary prior to orthodontic treatment. Angle Orthod. 2010 Mar;80(2):262-6. doi: 10.2319/111608-588.1. PMID 19905850
- [Result] Turakhia MP, Desai M, Hedlin H, Rajmane A, Talati N, Ferris T, Desai S, Nag D, Patel M, Kowey P, Rumsfeld JS, Russo AM, Hills MT, Granger CB, Mahaffey KW, Perez MV. Rationale and design of a large-scale, app-based study to identify cardiac arrhythmias using a smartwatch: The Apple Heart Study. Am Heart J. 2019 Jan;207:66-75. doi: 10.1016/j.ahj.2018.09.002. Epub 2018 Sep 8. PMID 30392584
- [Result] Topalovic M, Das N, Burgel PR, Daenen M, Derom E, Haenebalcke C, Janssen R, Kerstjens HAM, Liistro G, Louis R, Ninane V, Pison C, Schlesser M, Vercauter P, Vogelmeier CF, Wouters E, Wynants J, Janssens W; Pulmonary Function Study Investigators; Pulmonary Function Study Investigators:. Artificial intelligence outperforms pulmonologists in the interpretation of pulmonary function tests. Eur Respir J. 2019 Apr 11;53(4):1801660. doi: 10.1183/13993003.01660-2018. Print 2019 Apr. PMID 30765505
- [Result] Thanathornwong B. Bayesian-Based Decision Support System for Assessing the Needs for Orthodontic Treatment. Healthc Inform Res. 2018 Jan;24(1):22-28. doi: 10.4258/hir.2018.24.1.22. Epub 2018 Jan 31. PMID 29503749
- [Result] Suhail Y, Upadhyay M, Chhibber A, Kshitiz. Machine Learning for the Diagnosis of Orthodontic Extractions: A Computational Analysis Using Ensemble Learning. Bioengineering (Basel). 2020 Jun 12;7(2):55. doi: 10.3390/bioengineering7020055. PMID 32545428
- [Result] Lee JH, Kim DH, Jeong SN, Choi SH. Detection and diagnosis of dental caries using a deep learning-based convolutional neural network algorithm. J Dent. 2018 Oct;77:106-111. doi: 10.1016/j.jdent.2018.07.015. Epub 2018 Jul 26. PMID 30056118
- [Result] Lee KS, Jung SK, Ryu JJ, Shin SW, Choi J. Evaluation of Transfer Learning with Deep Convolutional Neural Networks for Screening Osteoporosis in Dental Panoramic Radiographs. J Clin Med. 2020 Feb 1;9(2):392. doi: 10.3390/jcm9020392. PMID 32024114
- [Result] Skotko BG, Macklin EA, Muselli M, Voelz L, McDonough ME, Davidson E, Allareddy V, Jayaratne YS, Bruun R, Ching N, Weintraub G, Gozal D, Rosen D. A predictive model for obstructive sleep apnea and Down syndrome. Am J Med Genet A. 2017 Apr;173(4):889-896. doi: 10.1002/ajmg.a.38137. Epub 2017 Jan 26. PMID 28124477
- [Result] Patcas R, Timofte R, Volokitin A, Agustsson E, Eliades T, Eichenberger M, Bornstein MM. Facial attractiveness of cleft patients: a direct comparison between artificial-intelligence-based scoring and conventional rater groups. Eur J Orthod. 2019 Aug 8;41(4):428-433. doi: 10.1093/ejo/cjz007. PMID 30788496
- [Result] Patcas R, Bernini DAJ, Volokitin A, Agustsson E, Rothe R, Timofte R. Applying artificial intelligence to assess the impact of orthognathic treatment on facial attractiveness and estimated age. Int J Oral Maxillofac Surg. 2019 Jan;48(1):77-83. doi: 10.1016/j.ijom.2018.07.010. Epub 2018 Aug 4. PMID 30087062
- [Result] Li P, Kong D, Tang T, Su D, Yang P, Wang H, Zhao Z, Liu Y. Orthodontic Treatment Planning based on Artificial Neural Networks. Sci Rep. 2019 Feb 14;9(1):2037. doi: 10.1038/s41598-018-38439-w. PMID 30765756
- [Result] Ma Q, Kobayashi E, Fan B, Nakagawa K, Sakuma I, Masamune K, Suenaga H. Automatic 3D landmarking model using patch-based deep neural networks for CT image of oral and maxillofacial surgery. Int J Med Robot. 2020 Jun;16(3):e2093. doi: 10.1002/rcs.2093. Epub 2020 Mar 20. PMID 32065718
- [Result] Nino-Sandoval TC, Guevara Perez SV, Gonzalez FA, Jaque RA, Infante-Contreras C. Use of automated learning techniques for predicting mandibular morphology in skeletal class I, II and III. Forensic Sci Int. 2017 Dec;281:187.e1-187.e7. doi: 10.1016/j.forsciint.2017.10.004. Epub 2017 Oct 12. PMID 29126697
- [Result] Nieri M, Crescini A, Rotundo R, Baccetti T, Cortellini P, Pini Prato GP. Factors affecting the clinical approach to impacted maxillary canines: A Bayesian network analysis. Am J Orthod Dentofacial Orthop. 2010 Jun;137(6):755-62. doi: 10.1016/j.ajodo.2008.08.028. PMID 20685530
- [Result] Nanda, R. (2012) 'Biomechanics and Esthetics Strategies in Clinical Orthodontics', Paper Knowledge . Toward a Media History of Documents, p. 194.
- [Result] Nahidh, M., Am, A. A. and Sc, A. (2019) 'Understanding Anchorage in Orthodontics', ARC Journal of Dental Science, 4(3). doi: 10.20431/2456-0030.0403002.
- [Result] Montufar J, Romero M, Scougall-Vilchis RJ. Hybrid approach for automatic cephalometric landmark annotation on cone-beam computed tomography volumes. Am J Orthod Dentofacial Orthop. 2018 Jul;154(1):140-150. doi: 10.1016/j.ajodo.2017.08.028. PMID 29957312
- [Result] Mitchell, L. (2017) 'Introduction to Orthodontics', in Introduction to Orthodontics. 4th edn, pp. 179-190.
- [Result] Mendes RG, de Souza CR, Machado MN, Correa PR, Di Thommazo-Luporini L, Arena R, Myers J, Pizzolato EB, Borghi-Silva A. Predicting reintubation, prolonged mechanical ventilation and death in post-coronary artery bypass graft surgery: a comparison between artificial neural networks and logistic regression models. Arch Med Sci. 2015 Aug 12;11(4):756-63. doi: 10.5114/aoms.2015.48145. Epub 2015 Aug 11. PMID 26322087
- [Result] Martina, R. et al. (2006) 'Neural Network Based System for Decision Making Support in Orthodontic Extractions', Intelligent Production Machines and Systems - 2nd I*PROMS Virtual International Conference 3-14 July 2006, pp. 235-240. doi: 10.1016/B978-008045157-2/50045-6.
- See also: Related Info — http://www.amazon.com/001-Tips-Orthodontics-its-Secrets/dp/9381714398

DOCUMENTS (1):
  • Study Protocol (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT05348109/Prot_000.pdf